CLINICAL TRIAL: NCT01753492
Title: Trabeculectomy With Ologen-Pilot
Brief Title: Trabeculectomy With Ologen
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The results were disappointing.
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Aeon Astron Europe B.V. (Industry)
Responsible Party: Principal Investigator, Henny Beckers, MD, PhD, Ophthalmologist, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL42312.068.12/METC12-2-073
Record Dates: First submitted 2012-12-12; First posted 2012-12-20 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Glaucoma
Keywords: Intraocular pressure; glaucoma; trabeculectomy; Ologen
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ologen implantation (single arm) (Experimental): Ologen implantation as an adjunctive to trabeculectomy
  Interventions: Device: Ologen

INTERVENTIONS:
Device: Ologen

SUMMARY:
Trabeculectomy is the gold standard procedure for the surgical treatment of glaucoma. Antimetabolites such as mitomycin-C (MMC)are widely used as an adjunctive during surgery to prevent scarring of the bleb. MMC has the risk for creating thin bleb walls, avascular blebs, and increased risk to infection, blebitis and endophthalmitis.

Recently, a biodegradable porous collagen-glycosaminoglycan copolymer matrix implant (Ologen), has become available for glaucoma surgery.Although a few studies on filtering surgery with Ologen implantation have been performed, there is yet no conclusive evidence on effectivity and safety with Ologen implantation when compared to trabeculectomy with MMC.

This is a prospective intervention pilot study to determine the degree of intraocular pressure (IOP) lowering of trabeculectomy with Ologen implantation in comparison to trabeculectomy with MMC. Additionally, the safety (per- and postoperative complications) of the two procedures will be compared.

The study hypothesis is that trabeculectomy with Ologen will be a safer procedure than trabeculectomy with MMC, but probably at the cost of a less potent IOP lowering.

ELIGIBILITY:
Inclusion Criteria:

* Primary open-angle glaucoma with progression of visual field loss and/or uncontrolled intraocular pressure levels with medication.
* Indication for trabeculectomy with mitomycin-C

Exclusion Criteria:

* Unability to discontinue oral anticoagulants
* Difficulty in reading or speaking Dutch
* Previous ocular surgery (cataract surgery allowed)
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Postoperative intraocular pressure level | 3 months

SECONDARY OUTCOMES:
Number of glaucoma medications | 3 months

OTHER OUTCOMES:
bleb aspect: hyperemia (grade 1, 2 or 3), bleb height (1, 2 or 3) | 3 months
surgery time | 3 months
complexity of surgical procedure | 3 months
number of patients withdrawn from study because of failure | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Clinic, Maastricht, Netherlands